CLINICAL TRIAL: NCT05502965
Title: Effectiveness and Pathogenesis of Specific Dietary Pattern in Maintaining Remission Among Crohn's Disease(CD) Patients Following Surgery
Brief Title: Specific Dietary Pattern for Crohn's Disease Patients Following Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2022-0454
Record Dates: First submitted 2022-08-11; First posted 2022-08-16 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Crohn Disease
Keywords: Dietary Pattern, Crohn Disease
MeSH Terms: conditions — Crohn Disease | interventions — Dietary Patterns

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exclusive Enteral Nutrition(EEN) (Active Comparator): Subjects required exclusive enteral nutrition for one month
  Interventions: Other: EEN
- Specific Diet+ Partial Enteral Nutrition (Experimental): Subjects received partial enteral nutrition with remaining energy and nutrients obtained through diet for one month
  Interventions: Other: dietary pattern

INTERVENTIONS:
Other: dietary pattern — Reprocessed and intolerant foods were removed from the dietary pattern, and the food were cooked at home for experimental subjects.
  Other Names: dietary guidance
  Arms: Specific Diet+ Partial Enteral Nutrition
Other: EEN — All energy and nutrients are obtained from exclusive enteral nutrition.
  Arms: Exclusive Enteral Nutrition(EEN)

SUMMARY:
Over the past 10 years, there are a large number of dietary treatments related to the CD, such as specific carbohydrate diet, low Fermentable Oligo-, Di-, Mono-saccharides And Polyols (FODMAP) diet, and allergen-free foods. But there is no consistent conclusion or convincing evidence about the effectiveness. Through the long-term clinical experience observation, we find most of the CD patients can get stable remission by removing refined food and intolerance food.This project aims at developing a new dietary therapy suitable for Chinese patients.

DETAILED DESCRIPTION:
The dietary therapy is based on the nutrient composition of exclusive enteral nutrition and is more in line with Chinese patients' dietary habits and economic conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnose CD according to endoscopy, histology and imaging;
2. Bowel resection for CD
3. Oral nutritional preparations or food can be given after surgery

Exclusion Criteria:

1. Plan operation within 5 weeks after surgery;
2. Presence of an ileostomy or colostomy
3. Complete bowel obstruction or fibrous stricture
4. Pregnancy or breastfeeding;
5. Plan to use biological agents within 5 weeks after surgery;
6. Plan to use corticosteroids or prednisone greater than 20 mg per day or equivalent doses of drugs to maintain remission within 5 weeks after surgery;
7. Plan to use probiotics or prebiotics for more than 1 week after surgery;
8. Antibiotics are used for more than 2 weeks after surgery;
9. Hypersensitivity to known components of enteral nutrition;
10. BMI less than 14 or greater than 28 kg/m2;
11. Celiac disease;
12. Complicated with other autoimmune diseases such as diabetes or rheumatic disease, autoimmune liver disease, psoriasis;
13. Mental illness;
14. Malignant tumors
15. Those who are not suitable for body composition analysis (such as pacemakers and metal objects in the body)
16. Participating in other clinical trials
17. The researcher believes that others are not suitable to participate in this study.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2022-09-17 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Quality of Life(IBDQ) | The two groups of patients were scored at first week and sixth week after surgery.
  IBDQ: Inflammatory Bowel Disease Questionnaire.The IBDQ evaluates the quality of life of patients from four aspects: intestinal symptoms, systemic symptoms, emotional function and social function. There are 32 questions in the questionnaire, with a total score of 32 to 224 points. The higher the score, the higher the quality of life of the patient.

SECONDARY OUTCOMES:
nutritional status of the patient | The two groups were evaluated at first week and sixth week after surgery.
  Body composition analysis, calf circumference in centimeter , albumin in g/L, hemoglobin in g/L, were measured to evaluate the nutritional status
Disease-related evaluation indicators | The two groups were evaluated at first week and sixth week after surgery.
  We assessed the effect of the intervention on disease by measuring the following indicators: Harvey-Bradshaw Index(HBI), Crohn's Disease Activity Index (CDAI), C Reactive Protein (CRP)in mg/L, Erythrocyte Sedimentation Rate (ESR) in mm/h, platelets in 10^9/L, triglycerides in m mol/L, cholesterol in m mol/L , uric acid in u mol/L.

OTHER OUTCOMES:
dietary compliance | The two groups were evaluated at sixth week after surgery.
  Modified medication adherence was measured, with < 6 points defined as low adherence, 6 to 8 points defined as moderate adherence, and > 8 points defined as high adherence

CONTACTS AND LOCATIONS:
Overall Officials: yu qiao, Principal Investigator — 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China; guo huilan, Study Director — 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No